CLINICAL TRIAL: NCT05244135
Title: Implementation of an Innovative Hospital Pulmonary Rehabilitation Based on Virtual Reality for Post-COVID-19 Patients
Brief Title: Pulmonary Rehabilitation Implemented With Virtual Reality for Post-COVID-19 Patients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: The Opole University of Technology (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: COVID_2
Record Dates: First submitted 2022-02-15; First posted 2022-02-17 (Actual); Last update posted 2022-07-13 (Actual); Status verified 2022-07

CONDITIONS: COVID-19
Keywords: COVID-19; Pulmonary rehabilitation; Virtual Reality
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Pulmonary rehabilitation in VR (VR group) (Experimental): The VR group will perform the endurance exercise training using the "Virtual Park", developed by CNR-STIIMA. The system includes a COSMED cycle-ergometer, a virtual environment and a physiological sensor-either a HR band or a pulse-oximeter depending on the target patient's needs. The virtual environment represents a ride in a park, enriched with realistic elements and sound effects, in order to simulate a daily life situation.
  In the VR group, the VR Tier One device (Stolgraf®) will be used as a VR source. Thanks to using a head mounted display and the phenomenon of total immersion, VR therapy provides an intense visual, auditory and kinaesthetic stimulation. The aim of the software was to calm and improve the mood, while motivating and cognitively activating the patient.
  Interventions: Procedure: Pulmonary rehabilitation
- Traditional Pulmonary Rehabilitation (TPR) (Active Comparator): In the TPR group, exercise training will be performed on the bicycle. The training will be conducted on cycle ergometers with the use of the Peloton™ system, which ensures the monitoring of performance parameters.
  In the TPR group, Schultz Autogenous Training will be performed. Schultz Autogenic Training has been shown to be effective in treating these pathologies. In both groups the relaxation training will be carried out once a day and will last about 20 minutes.
  Interventions: Procedure: Pulmonary rehabilitation

INTERVENTIONS:
Procedure: Pulmonary rehabilitation — An in-patients 3-week high intensity rehabilitation program, five times a week, was used as the intervention treatment. A holistic pulmonary rehabilitation program for SARS-CoV-2 patients with combined treatment focused on increasing exercise capacity, restoring lung function, and supporting mental health, developed by a multidisciplinary team, was introduced. Rehabilitation program includes exercise capacity training on a cycle ergometer, breathing exercises, general fitness exercises, resistance training, and relaxation.

SUMMARY:
Over recent months, SARS-CoV-2 infection has been confirmed in millions of people around the world. Furthermore, the COVID-19 pandemic gives rise to new psychosocial and emotional stressors for recovering patients, including social isolation, physical distancing, loss of employment and uncertainties about the future. This project is aimed to propose an innovative comprehensive intervention based on a stationary pulmonary rehabilitation (PR) programme for COVID-19 survivors. Moreover, this project assumes the use of virtual reality (VR) in rehabilitation processes.

DETAILED DESCRIPTION:
COVID-19 caused by SARS-CoV-2 has led to a global public health crisis. Millions of people around the world are infected with a severe acute respiratory coronavirus, causing COVID-19. Some of the patients with confirmed COVID-19 are admitted to hospital for acute care due to severe respiratory symptoms and coronary artery disease and, in some cases, even acute respiratory symptoms requiring prolonged mechanical ventilation. It is highly anticipated that some patients with COVID-19 will have a need for rehabilitation interventions during and immediately after hospitalization. However, data on safety and efficacy of rehabilitation during and/or after hospitalization in these patients are lacking. The benefits of respiratory rehabilitation are well known and existing programmes can be used as one of the referral paths for the rehabilitation of COVID-19 survivors with symptoms and/or impairment of physical functions. Many scrutinies and systematic literature reviews show the beneficial effect of pulmonary rehabilitation in patients with chronic respiratory diseases on exercise capacity, lung function, respiratory muscle strength, quality of life. Therefore, we assumed that the mechanisms leading to improvement of the psychosomatic condition will be the same as those in COVID-19 survivors because they present with the same clinical symptoms. This project is aimed to propose an innovative comprehensive intervention based on a stationary pulmonary rehabilitation (PR) programme for COVID-19 survivors. In our project, we intend to answer the following questions:

1. Whether participation in the 3-week pulmonary rehabilitation programme will change the pulmonary function and exercise capacity of individuals after infection with SARS-CoV-2?
2. Whether participation in the 3-week pulmonary rehabilitation programme will change the mental condition of individuals after infection with SARS-CoV-2 ?
3. Whether the implementation of immersive VR therapy in a pulmonary rehabilitation programme for post-COVID-19 patients will change the effectiveness compared to the traditional form of rehabilitation?

ELIGIBILITY:
Inclusion Criteria:

* Women and men aged 40-60 years who were hospitalized for COVID-19.

Exclusion Criteria:

* No consent to participate,
* active pneumonia diagnosed by x-ray,
* documented heart disease (stable or unstable),
* status after CABG, PTCA,
* uncontrolled hypertension,
* insulin-dependent diabetes mellitus,
* inability to exercise independently or musculoskeletal/neurological conditions that would prevent completion of the course,
* lung cancer,
* cognitive impairment or Mini-Mental State Examination < 24.

Ages: 40 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 66 (Estimated)
Dates: Start 2022-02-28 (Actual); Primary Completion 2022-03-21 (Actual); Study Completion 2022-09-30 (Estimated)

PRIMARY OUTCOMES:
Lung function | 10 minutes
  Spirometry testing will be performed in all patients before and after rehabilitation. For the assessment of respiratory function, the following indicators will be used: forced vital capacity (FVC), forced expiratory volume in one second (FEV1), and FEV1 percentage obtained the current VC (FEV1%). The measurement will be performed three times by the patient and the best result will be included in the research study.
Dyspnea | 2 minutes
  In all patients, prior to and immediately after the 6-minute walk test, an assessment of dyspnoea will be made by the 10-degree Borg scale, which is the most versatile and most widely used scale for breathlessness. This method will allow for comparison of the absolute level of breathlessness patients feel at a given exercise intensity. A lower score means less impairment
Stress | 5 minutes
  The Perceived Stress Scale (PSS) is the most widely used psychological instrument for measuring the perception of stress. It is a measure of the degree to which situations in one's life are appraised as stressful. Items were designed to tap how unpredictable, uncontrollable, and overloaded respondents find their lives. The scale also includes a number of direct queries about current levels of experienced stress. A lower score means less impairment
Anxiety and depression | 5 minutes
  The HADS is a 14-item scale, scoring each item from 0 to 3. The first seven items relate to anxiety (HADS-A), and the remaining seven items relate to depression (HADS-D). The global scoring ranges from 0 to 42, with a cut-off point of 8/21 for anxiety and 8/21 for depression. The higher the score is, the greater the anxiety or depression symptoms. The scale is considered to be a valid research method.
Individual's perception of quality of life | 10 minutes
  The WHO Quality of Life-BREF questionnaire is designed to assess the quality of life of healthy and sick people, both for cognitive and clinical purposes. It contains 26 questions analysing four areas of life: physical, psychological, social and environmental. A lower score means a poorer quality of life

SECONDARY OUTCOMES:
Heart Rate Variability | 30 minutes
  During trainings, Polar H10 monitor (Polar Electro Oy Inc., Kempele, Finland) will be employed to record HR series at a sampling frequency of 1000 Hz. The device is recommended as the gold standard for R-R interval assessments during intense activities to obtain HR and HRV. All HRV analyses will be carried out with the Kubios HRV Premium version 3.3.1
Impact of technology | 10 minutes
  The following scales will be used to evaluate immersive VR technology:
  System Usability (immersive VR group): System Usability Scale (SUS) Cyber illness (immersive VR group): Simulator Sickness Questionnaire (SSQ) Anxiety/negative affect (while using VR): the Positive and Negative Affect Scale (PANAS)

CONTACTS AND LOCATIONS:
Locations (1):
- MSWiA Specialist Hospital in Głuchołazy, Głuchołazy, Opole Voivodeship, Poland

IPD SHARING:
Plan to Share IPD: Undecided
Undecided

REFERENCES:
- [Derived] Rutkowski S, Bogacz K, Czech O, Rutkowska A, Szczegielniak J. Effectiveness of an Inpatient Virtual Reality-Based Pulmonary Rehabilitation Program among COVID-19 Patients on Symptoms of Anxiety, Depression and Quality of Life: Preliminary Results from a Randomized Controlled Trial. Int J Environ Res Public Health. 2022 Dec 17;19(24):16980. doi: 10.3390/ijerph192416980. PMID 36554860